CLINICAL TRIAL: NCT02788032
Title: Open Label Study of Acceptability, Tolerance, and Compliance Using EnergieShake® Dietary Powdered Supplement
Brief Title: EnergieShake® Acceptability and Tolerance Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anaiah Healthcare Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AHCES 005
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EnergieShake Intervention (Other): Single arm of intervention of Oral Nutritional Supplement in the open label study to be given to participants for 8 days Two 57g sachets of EnergieShake daily to be given to participants during the 8 day intervention period.
  Interventions: Other: EnergieShake oral supplement

INTERVENTIONS:
Other: EnergieShake oral supplement — The participants will be given EnergieShake® powdered nutritional supplement twice daily during the study period in place of their usual ONS. Participants will take their usual ONS for 2 days followed by an 8 day intervention on EnergieShake®

SUMMARY:
This open-label, prospective, controlled intervention study involves evaluating tolerance and acceptability of an Oral Nutrition Supplement (ONS; EnergieShake®) in 16 adult patients who are already taking an ONS. Following a 2-day baseline data collection on their current ONS, patients switch to the test ONS, which is taken for a further 8 consecutive days. Patients revert to their current ONS at the end of the study. Patients act as their own controls and thus all patients are allocated the same intervention.

Daily records of GI tolerance and compliance with the prescribed amount of ONS will be kept for participants throughout the study period. Participants' height and weight will be collected at baseline (weight at end will also be collected), all medications will be documented, and relevant medical and dietary histories will be recorded. A questionnaire at the end of the intervention period will be administered collecting participants' views on the acceptability (taste and palatability) of the test ONS. Taste and palatability will be assessed via a questionnaire that uses a Hedonic scale to quantify preference.

DETAILED DESCRIPTION:
INTRODUCTION, BACKGROUND INFORMATION AND SCIENTIFIC RATIONALE

Background Information

This open-label study involves evaluating tolerance and acceptability of the test ONS in 16 adult participants who are already taking an ONS. Following a 2-day baseline data collection on their current ONS, patients switch to the test ONS, which is taken for a further 8 consecutive days. Patients revert to their current ONS at the end of the study. Patients act as their own controls and thus all patients are allocated the same intervention.

Rationale

Patient tolerance and acceptability is fundamental to the successful use of an ONS. Acceptability and tolerance studies for ONS are required by the Advisory Committee on Borderline Substances (ACBS) as part of a submission for a new product to be made available at NHS expense in the community.

Potential Risks and Benefits

Potential Risks

There are no anticipated risks to participants. Participants will already be taking other ONS as this is one of the inclusion criteria. Minimal inconvenience to participants is anticipated as they will be asked to complete a questionnaire on the product's acceptability. Daily records on the GI tolerance of the product will be recorded by participants or nursing staff. Most of the study documentation will be completed by the study staff.

Potential Benefits

Participants may gain weight or maintain their weight during the intervention. In the future, if this product becomes available on prescription, a wider variety of ONS available to patients may lessen taste fatigue associated with taking the same supplements over an extended period.

STUDY OBJECTIVES

Primary study objective

The primary objective of the study is to assess gastrointestinal (GI) tolerance (bowel frequency and consistency using the Bristol Stool Chart, nausea, vomiting, abdominal discomfort, wind, burping, flatulence) to a Test Oral Nutrition Supplement (EnergieShake®, a powdered nutritional supplement, classified as a Food for Special Medical Purposes for the dietary management of disease-related malnutrition) in patients requiring ONS.

Secondary study objective

The secondary objective is to assess acceptability of the product.

STUDY DESIGN

This study is an open-label, prospective, controlled intervention in which participants act as their own controls. Guidance from ACBS requires that acceptability and tolerance studies must normally be carried out on at least 15 patients in the intended target group for a period of 1 week. The design of this study has been based on the guidance provided by ACBS.

STUDY ENROLLMENT AND WITHDRAWAL

Strategies for Recruitment and Retention

Potentially suitable participants will be identified by staff at the site. Participants who may be suitable are those who are currently taking ONS and whose requirement for ONS is expected to continue for at least a further 2 weeks. They will be approached by staff at the site and provided with a Participant Information Sheet and letter of invitation from the sponsor (Anaiah Healthcare Ltd). To ensure this process is free from undue influence, residents will not be coerced or offered inducements to participate.

Subject Withdrawal

Reasons for Withdrawal

Participants will have the choice of whether or not to withdraw from the study at any stage for any reason. Should the participant experience any adverse event or discomfort due to consuming the product, the participant will be advised to stop using the product.

Handling of Subject Withdrawals or Subject Discontinuation of Study Intervention

If the participant discontinues the study before the intervention is complete, their permission will be sought to use the data collected on the use of the product. A replacement of a participant who withdraws will be recruited to meet the requirement target that at least 15 patients provide data on the test ONS.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* Participants with or at risk of malnutrition who are already taking ONS on a daily basis
* Participants expected to continue to require ONS for at least a further 2 weeks
* Participants able to give their informed consent to participate

Exclusion Criteria:

* Requirement of tube or parenteral nutrition.
* Participants receiving palliative care.
* Participants with chronic renal disease or liver failure.
* Participants requiring a milk/lactose free diet
* Participants with significant on-going gastrointestinal symptoms.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Tolerance: how well the participant tolerates the Oral Nutritional Supplement, including changes to gastrointestinal symptoms. | 10 days
  The primary objective of the study is to assess gastrointestinal (GI) tolerance (bowel frequency and consistency using the Bristol Stool Chart, nausea, vomiting, abdominal discomfort, wind, burping, flatulence) to test Oral Nutrition Supplement (EnergieShake®, a powdered nutritional supplement, classified as a Food for Special Medical Purposes for the dietary management of disease-related malnutrition) in patients requiring ONS.

SECONDARY OUTCOMES:
How acceptable the Oral Nutritional Supplement is to the participant, (taste, texture, aroma, consistency, etc.) Compliance with Oral Nutritional Supplement. | 10 days
  Assessment on Taste Questionnaire used asks patients to rate appearance, taste/flavour, texture/consistency, Aroma/smell, Taste/sweetness, and overall acceptability using Hedonic scale: 9 (like extremely) to 1 (dislike extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rodrigues, Masters, Principal Investigator — Anaiah Healthcare Ltd
Locations (1):
- Fermoyle Nursing Home, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No